CLINICAL TRIAL: NCT01011530
Title: A Phase I, Open-Label, Dose Escalation Study of MLN4924, a Novel Inhibitor of Nedd8-Activating Enzyme, in Adult Patients With Melanoma
Brief Title: Dose Escalation Study of MLN4924 in Adults With Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C15005
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — pevonedistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MLN4924 (Experimental): MLN4924 via IV infusion
  Interventions: Drug: MLN4924

INTERVENTIONS:
Drug: MLN4924 — Patients will be administered MLN4924 via an IV infusion. Each 21-day treatment cycle is composed of 2 weeks intermittent dosing of MLN4924 on Days 1, 4, 8 and 11, followed by a rest period of 10 days. A cohort of patients will receive a reduced first dose on Day 1, approximately half the strength of the dose received on Days 4, 8, 11 and dose will not be administered on Day 4 if the Day 1 dose is not tolerated.(Schedule A ramp-up), or continuous weekly dosing (Days 1, 8, and 15) of MLN4924 (Schedule B)

SUMMARY:
This is an open-label, multicenter, phase 1, dose escalation study that will evaluate the safety profile, establish Maximum Tolerated Dose (MTD), and inform the recommended phase 2 dose of MLN4924 as well as evaluate antitumor activity in patients with metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following criteria to be enrolled in the study:

* Diagnosis of metastatic melanoma
* Measurable disease
* Female patients who are post menopausal, surgically sterile, or agree to practice 2 effective methods of contraception or abstain from heterosexual intercourse
* Male patients who agree to practice effective barrier contraception or agree to abstain from heterosexual intercourse
* Willing and able to give written informed consent
* Suitable venous access for study-required blood sampling
* Appropriate functional status, including the recovery from the effects of prior antineoplastic therapy, and acceptable organ function as described in the protocol

Exclusion Criteria:

Patients meeting any of the following exclusion criteria are not to be enrolled in the study:

* Major surgery or, serious infections, or infections that required systematic antibiotic therapy within 14 days before the first dose of study drug
* Systemic antineoplastic or radiation therapy within 14 days or treatment with any investigational products within 21 days before the first dose of study treatment
* CYP3A inducers within 14 days of study treatment. Moderate and strong CYP3A inhibitors and CYP3A inducers are not permitted during the study
* No prior history of amiodarone in the 6 months before the first dose of MLN4924
* Diarrhea that is greater than Grade 1 as outlined in the protocol
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months
* Known human immunodeficiency virus (HIV) positive, hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection.
* Serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to the protocol
* Other clinical and laboratory assessments that do not meet the criteria specified in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-12; Primary Completion 2012-05 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) and inform recommended phase 2 dose of MLN4924 | Up to 12 months of treatment

SECONDARY OUTCOMES:
Anti-tumor activities of MLN4924 | Up to 12 months of treatment
Pharmacodynamic effects of MLN4924 on blood and tumor cells | Primarily assessed during the first cycle of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- The Angeles Clinic and Research Institute, Santa Monica, California, United States

REFERENCES:
- [Derived] Faessel HM, Mould DR, Zhou X, Faller DV, Sedarati F, Venkatakrishnan K. Population pharmacokinetics of pevonedistat alone or in combination with standard of care in patients with solid tumours or haematological malignancies. Br J Clin Pharmacol. 2019 Nov;85(11):2568-2579. doi: 10.1111/bcp.14078. Epub 2019 Sep 4. PMID 31355467